CLINICAL TRIAL: NCT07348094
Title: Computer-Guided Lateral Sinus Floor Elevation Using Autologous Serum Albumin/Platelet Rich Fibrin Combined With Serum Albumin Membrane: A Randomized Clinical Study
Brief Title: Guided Lateral Sinus Lifting Using Autologous Serum Albumin/Platelet-Rich Fibrin
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Walid Elamrousy, Professor of Periodontology Department Faculty of Oral and Dental Medicine,Kafrelsheikh University, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KFSIRB200-333
Record Dates: First submitted 2026-01-09; First posted 2026-01-16 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Sinus Perforation; Dental Implant Failure Nos
MeSH Terms: interventions — Bone Transplantation

STUDY DESIGN:
Intervention Model Description: guided Lateral sinus lift with bone graft only
Who Masked: Outcomes Assessor
Masking Description: outcome assessor is masked
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I (Experimental): Lateral window was done using surgical guide for placement of implants in posterior edentulous maxillary regions. Then bone graft only will be used.
  Interventions: Procedure: Guided Lateral Sinus Lifting with bone graft
- Group II (Experimental): Lateral window was done using surgical guide for placement of fifteen implants in posterior edentulous maxillary regions. Then an autologous Alb-PRF only will be used
  Interventions: Procedure: Guided Lateral Sinus Lifting with Autologous Serum Albumin/Platelet-Rich Fibrin
- Group III (Experimental): Lateral window was done using surgical guide for placement of fifteen implants in posterior edentulous maxillary regions. Then sticky bone [bone graft with Alb-PRF] only will be used
  Interventions: Procedure: Guided Lateral Sinus Lifting with sticky bone

INTERVENTIONS:
Procedure: Guided Lateral Sinus Lifting with bone graft — Lateral window was done using surgical guide for placement of fifteen implants in posterior edentulous maxillary regions. Then bone graft only will be used.
  Arms: Group I
Procedure: Guided Lateral Sinus Lifting with Autologous Serum Albumin/Platelet-Rich Fibrin — Lateral window was done using surgical guide for placement of fifteen implants in posterior edentulous maxillary regions. Then an autologous Alb-PRF only will be used
  Arms: Group II
Procedure: Guided Lateral Sinus Lifting with sticky bone — Lateral window was done using surgical guide for placement of fifteen implants in posterior edentulous maxillary regions. Then sticky bone [bone graft with Alb-PRF] only will be used
  Arms: Group III

SUMMARY:
This research aimed to evaluate the effect of an autologous Alb-PRF on bone regeneration after lateral sinus lifting via 3D volumetric analysis. The null hypothesis of this research was that there would be no significant difference between the group that would be treated by lateral sinus lift and Alb-PRF application and that would be treated by lateral sinus lift with bone graft for bone regeneration.

DETAILED DESCRIPTION:
Sinus floor augmentation became a widely accepted surgical procedure to improve the amount of bone volume before implant placement. According to the guided bone regeneration principles, in the sinus lift procedure, bone graft was demonstrated to act as space holder under the elevated sinus membrane. The osteogenic source for the bone healing derives from two different anatomic sites: the basal bone of the sinus cavity and the periosteum represented as basal cell layer of the Schneiderian membrane.

Proper and accurate design and location of the lateral side window is necessary to facilitate the sinus lifting process and help the surgeon to successfully lift the sinus membrane. In addition, direct visualization helps in better packing of the entire graft space, which is essential to provide primary stability for the simultaneous insertion of the implants with the sinus elevation procedure.

The application of digital technology has proven to be a valuable tool for diagnosis and treatment planning. Data obtained from CBCT scans, digital oral scans, and facial scans can be integrated and manipulated using special computer software, providing surgeons with an interactive interface to perform virtual surgery planning before the actual surgery.

The precision of stereolithographic guides may mitigate risks associated with anatomical variations in atrophic maxillae, potentially reducing membrane perforation and optimizing lateral window osteotomy and implant placement accuracy which are key factors this study evaluates.

Recently, the use of pure autologous concentrations of platelets, PRF, as a graft material has shown promising effects. However, the durability of PRF is limited, as it usually resorbs within 10-14 days. Thus, Mourão et al. introduced a new technique for PRF preparation, in which the resulting newly formed protein remains stable for a long time, up to 4 to 6 months. The buffy coat layer of the PRF was then mixed with the denatured albumin gel and cooled to room temperature to form a new autologous albumin gel-platelet-rich fibrin mixture (Alb-PRF) which has the ability to heal, represented by the delayed and gradual release of growth factors present in the buffy coat layer of PRF throughout the prolonged dissolution of the albumin gel.

This research aimed to evaluate the effect of an autologous Alb-PRF on bone regeneration after lateral sinus lifting via 3D volumetric analysis. The null hypothesis of this research was that there would be no significant difference between the group that would be treated by lateral sinus lift and Alb-PRF application and that would be treated by lateral sinus lift with bone graft for bone regeneration.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ≥18 years of age.

  * ASA I and ASA II.
  * Patients having partial edentulism in the posterior region of the maxilla.
  * Edentulous sites consist of native non augmented bone.
  * Horizontal ridge dimension minimum of 5mm
  * The vertical ridge dimension 3-6 mm.
  * Bone quality of D2 or D3.
  * Enough inter-arch distance.

Exclusion Criteria:

* - Patients with uncontrolled systemic diseases.
* History of chronic maxillary sinus pathology.
* Heavy smokers or patients with poor oral hygiene.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2027-01-30 (Estimated); Study Completion 2027-02-15 (Estimated)

PRIMARY OUTCOMES:
Implant stability | 12-months
  using implant stability quotient device

SECONDARY OUTCOMES:
Vertical bone height gain | 12 months
  assessed by CBCT.by measuring the distance from alveolar crest to sinus floor

IPD SHARING:
Plan to Share IPD: No